CLINICAL TRIAL: NCT05419128
Title: Family-focused vs. Drinker-focused Smartphone Interventions to Reduce Drinking-related Consequences of COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021-0943; 5R01AA029804 (NIH)
Record Dates: First submitted 2022-06-13; First posted 2022-06-15 (Actual); Results first posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Alcohol Use Disorder; Family Members; Behavior, Addictive
Keywords: mobile phone applications; quality of life; Alcohol Use Disorder; family therapy; high-risk drinking; alcohol behavioral couple therapy; COVID-19; mHealth; eHealth; ACHESS; PartnerCHESS
MeSH Terms: conditions — Alcoholism; Behavior, Addictive; COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ACHESS (Active Comparator): In ACHESS, both the identified patient and the concerned significant other will receive a smartphone, but only the identified patient will receive the ACHESS app. The concerned significant other will receive a smartphone with contact information for standard AUD, SUD, and crisis support.
  Interventions: Behavioral: ACHESS
- PartnerCHESS (Experimental): In the PartnerCHESS arm, identified patient and concerned significant other will both receive a smartphone with the PartnerCHESS app, which contains ACHESS services plus ABCT/ PartnerCHESS services.
  Interventions: Behavioral: PartnerCHESS
- Smartphone Control (No Intervention): Both the identified patient and concerned significant other will receive a smartphone with pre-programmed contact information for Alcoholics Anonymous (AA), Narcotics Anonymous (NA), Al-Anon, Adult Children of Alcoholics (ACOA), and crisis hot lines.

INTERVENTIONS:
Behavioral: PartnerCHESS — The following ABCT services, from PartnerCHESS, will be available in the PartnerCHESS app but not in ACHESS:
  ABCT tutorials. Interactive e-learning modules explaining key ABCT skills. Agreements between identified patient and concerned significant other to follow key principles.
  Trigger identification and removal. Cravings discussion. Relapse plan. Reminders.
  Arms: PartnerCHESS
Behavioral: ACHESS — ACHESS offers the following, which are also available in PartnerCHESS: Covid content, Instant Library, Discussion Groups, Personal Stories, Location Monitor, Surveys and Ecological Momentary Assessments, Guided Relaxation, Healthy Activities, Crisis Button, Skills Reminders
  Arms: ACHESS

SUMMARY:
This R01 project titled "Family-focused vs. Drinker-focused Smartphone Interventions to Reduce Drinking-related Consequences of COVID-19" is a Hybrid II RCT/implementation study to modify and test two of our alcohol smartphone interventions to address the fallout from COVID. We propose a three-arm RCT comparing a smartphone control group vs. a drinker-focused intervention vs. a family-focused intervention. All study arms recruit dyads comprising a person who drinks and a family partner.

DETAILED DESCRIPTION:
The current randomized controlled trial tested whether PartnerCHESS (an ACHESS intervention along with aspects of Alcohol Behavioral Couple Therapy designed specifically for individuals with alcohol use disorder and their concerned significant other) could reduce high-risk drinking and improve quality of life.

For this trial, 199 dyads (398 participants) were recruited from the community and randomized 1:1:1 to the PartnerCHESS intervention, ACHESS intervention, or smartphone control for 8 months with a follow-up at 12 months. Participants were part of a dyad: identified patients met criteria for high-risk drinking (defined by the DSM-5) and had at least one drink in the past month, concerned significant others were the identified patient's romantic partner, family member, or close friend aged 21 or older. Primary outcomes were identified patient percent high-risk drinking days, and quality of life for both identified patients and concerned significant others. Participants were surveyed at baseline, 4, 8, and 12 months; PartnerCHESS and ACHESS usage data were continuously collected. We found significant difference in both PartnerCHESS and ACHESS arms compared to smartphone control in percent high-risk drinking days as well as identified patient quality of life. Additionally, PartnerCHESS had significantly lower percent high-risk drinking days than ACHESS at 12 months, suggesting a stronger long-term impact. We also found significantly less distress among ACHESS concerned significant others as compared to those in PartnerCHESS and the smartphone control arms.

ELIGIBILITY:
Inclusion Criteria:

* Identified patients and their concerned significant others must give informed consent; agree to complete interviews at baseline, 4, 8, and 12 months; and not have a mental or physical condition that limits smartphone use. Identified patients must be age 18 or older and meet criteria for risky drinking (for men, >4 standard drinks in a day; for women, >3 in a day), or meet criteria for AUD (any severity) defined by DSM-5 and have had at least 1 drink in the past 3 months . Partner must be a committed romantic partner/spouse, close friend or family member (e.g. sibling, parent, grandparent, adult child age 21 or older).

Exclusion Criteria:

* Individuals were not eligible if they had current (last 6 months) evidence of serious mental illness (eg, active psychosis, active manic phase), or if either partner reported serious interpersonal violence, to avoid risk of violence from engagement on potentially sensitive subjects.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 398 (Actual)
Dates: Start 2022-04-06 (Actual); Primary Completion 2024-07-02 (Actual); Study Completion 2024-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Gustafson, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was conducted from April 2022 to May 2023. The intervention period ended in June 2024.
Pre-assignment Details: No significant events occurred after enrollment and prior to assignment.
Groups:
- Smartphone Control - Identified Patient (IP); Smartphone Control - Concerned Significant Other (CSO): Both the identified patient (IP) and concerned significant other (CSO) will receive a smartphone with pre-programmed contact information for Alcoholics Anonymous (AA), Narcotics Anonymous (NA), Al-Anon, Adult Children of Alcoholics (ACOA), and crisis hot lines.
- ACHESS - Identified Patient (IP); ACHESS - Concerned Significant Other (CSO): In ACHESS, both the identified patient (IP) and the concerned significant other (CSO) will receive a smartphone, but only the IP will receive the ACHESS app. The CSO will receive a smartphone with contact information for standard AUD, SUD, and crisis support.
  ACHESS: ACHESS offers the following, which are also available in PartnerCHESS: Covid content, Instant Library, Discussion Groups, Personal Stories, Location Monitor, Surveys and Ecological Momentary Assessments, Guided Relaxation, Healthy Activities, Crisis Button, Skills Reminders
- PartnerCHESS - Identified Patient (IP); PartnerCHESS - Concerned Significant Other (CSO): In the PartnerCHESS arm, identified patient (IP) and concerned significant other (CSO) will both receive a smartphone with the PartnerCHESS app, which contains ACHESS services plus ABCT/ PartnerCHESS services.
  PartnerCHESS: The following ABCT services, from PartnerCHESS, will be available in the PartnerCHESS app but not in ACHESS:
  ABCT tutorials. Interactive e-learning modules explaining key ABCT skills. Agreements between IP and CSO to follow key principles. Trigger identification and removal. Cravings discussion. Relapse plan. Reminders.
Period: Overall Study
Arm/Group | Smartphone Control - Identified Patient (IP) | ACHESS - Identified Patient (IP) | PartnerCHESS - Identified Patient (IP) | Smartphone Control - Concerned Significant Other (CSO) | ACHESS - Concerned Significant Other (CSO) | PartnerCHESS - Concerned Significant Other (CSO)
Started | 67 | 66 | 66 | 67 | 66 | 66
Completed | 66 | 65 | 65 | 66 | 65 | 65
Not Completed | 1 | 1 | 1 | 1 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Smartphone Control - Identified Patient (IP) | ACHESS - Identified Patient (IP) | PartnerCHESS - Identified Patient (IP) | Smartphone Control - Concerned Significant Other (CSO) | ACHESS - Concerned Significant Other (CSO) | PartnerCHESS - Concerned Significant Other (CSO) | Total
Number analyzed (Participants) | 67 | 66 | 66 | 67 | 66 | 66 | 398
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.0 (13.2) | 46.5 (13.3) | 46.4 (13.4) | 49.5 (13.2) | 48.5 (16.0) | 46.2 (14.3) | 47.5 (14.0)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Man, Woman, or Other (nonbinary, prefer not to say, etc.)
  Participants
    Man | 40 | 38 | 41 | 19 | 23 | 15 | 176
    Woman | 25 | 28 | 25 | 48 | 42 | 51 | 219
    Other | 2 | 0 | 0 | 0 | 1 | 0 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 6 | 7 | 2 | 4 | 6 | 28
  Not Hispanic or Latino | 63 | 60 | 59 | 65 | 62 | 60 | 369
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Percentages do not sum to 100 because participants could endorse multiple times.
  Participants
    White | 52 | 50 | 53 | 55 | 51 | 54 | 315
    African American | 11 | 13 | 9 | 10 | 11 | 8 | 62
    Other | 6 | 6 | 7 | 3 | 7 | 7 | 36
    Unknown | 1 | 0 | 0 | 0 | 0 | 0 | 1
Living arrangement [Count of Participants; unit: Participants] — Percentages do not sum to 100 because participants could endorse multiple times.
  Participants
    By myself | 14 | 14 | 10 | 8 | 6 | 10 | 62
    With a romantic partner | 42 | 38 | 36 | 50 | 48 | 38 | 252
    Other | 27 | 27 | 32 | 25 | 28 | 31 | 170
    Unknown | 1 | 0 | 0 | 0 | 0 | 0 | 1
Dyad relationship type [Count of Participants; unit: Participants] — Relationship type based on survey at baseline (some dyads had a discrepancy on how they defined their relationship, for example: romantic vs. friend).
  Participants
    Romantic partner/spouse | 44 | 43 | 39 | 45 | 43 | 38 | 252
    Parent/adult child/other family member | 15 | 18 | 23 | 15 | 18 | 23 | 112
    Friend | 8 | 5 | 4 | 7 | 5 | 5 | 34
Employment status [Count of Participants; unit: Participants] — Percentages do not sum to 100 because participants could endorse multiple times.
  Participants
    Employed full time | 25 | 37 | 28 | 37 | 31 | 32 | 190
    Employed part time/seasonal/other | 15 | 5 | 9 | 15 | 9 | 13 | 66
    Looking for work | 11 | 10 | 10 | 2 | 7 | 7 | 47
    On disability | 9 | 9 | 4 | 6 | 5 | 4 | 37
    Other | 10 | 8 | 15 | 8 | 14 | 11 | 66
    Unknown | 1 | 0 | 0 | 0 | 0 | 0 | 1
Vaccinated for COVID [Count of Participants; unit: Participants]
  Vaccinated for COVID | 47 | 49 | 46 | 53 | 51 | 49 | 295
  Unknown | 1 | 0 | 0 | 0 | 0 | 0 | 1
Past month drug use or abuse [Count of Participants; unit: Participants] — Percentages do not sum to 100 because participants could endorse multiple times.
  Participants
    Opioids/Sedatives/Tranquilizers | 2 | 2 | 4 | 4 | 2 | 2 | 16
    Marijuana | 28 | 21 | 28 | 9 | 13 | 15 | 114
    Stimulants | 5 | 5 | 5 | 1 | 2 | 3 | 21
    Unknown | 1 | 0 | 0 | 0 | 0 | 0 | 1
Past month treatment [Count of Participants; unit: Participants] — Percentages do not sum to 100 because participants could endorse multiple times.
  Participants
    Past month treatment | 16 | 19 | 21 | 1 | 9 | 4 | 70
    No past month treatment | 50 | 47 | 45 | 66 | 57 | 62 | 327
    Unknown | 1 | 0 | 0 | 0 | 0 | 0 | 1
Past month treatment engagement [Count of Participants; unit: Participants] — Percentages do not sum to 100 because participants could endorse multiple times.
  Participants
    Outpatient treatment | 6 | 11 | 14 | 0 | 6 | 3 | 40
    Inpatient treatment | 11 | 12 | 9 | 1 | 3 | 1 | 37
    Medically Assisted Treatment (MAT) use | 11 | 10 | 12 | 0 | 4 | 3 | 40
    Unknown | 1 | 0 | 0 | 0 | 0 | 0 | 1
Other healthcare utilization [Count of Participants; unit: Participants] — Percentages do not sum to 100 because participants could endorse multiple times.
  12-step/self-help group could include Al-Anon. meetings. Emergency room visit reasons were not specified.
  Participants
    12-step/self-help group | 12 | 20 | 15 | 5 | 13 | 7 | 72
    Emergency room visit | 12 | 11 | 6 | 5 | 3 | 3 | 40
    Unknown | 1 | 0 | 0 | 0 | 0 | 0 | 1
Severe Alcohol Use Disorder [Count of Participants; unit: Participants] — Based on DSM-5, Mild is defined as having 2-3 symptoms, Moderate is defined as having 4-5 symptoms, Severe is defined as having 6 or more symptoms (out of 11 total), only Identified Patients were screened for Alcohol Use Disorder eligibility. Population: Only Severe Alcohol Use was calculated, participants not shown had mild or moderate Alcohol Use Disorder as determined by the DSM-5.
  Participants
    number analyzed (Participants) | 67 | 66 | 66 | 0 | 0 | 0 | 199
    (all) | 62 | 65 | 59 |  |  |  | 186

OUTCOME MEASURES:

1. Primary Outcome: % of Patient Risky Drinking Days
Description: Risky drinking day will be defined as greater than 4 drinks for men and greater than 3 drinks for women and will be measured through the Timeline Followback every 120 days.
Time Frame: Baseline, 4, 8, and 12 months
Population: Identified Patients in each arm (Smartphone Control, ACHESS, and PartnerCHESS) were surveyed at baseline, 4, 8, and 12 months.
Measure: Mean (Standard Error); unit: percentage of high-risk drinking days
Arm/Group | Smartphone Control - Identified Patient (IP) | ACHESS - Identified Patient (IP) | PartnerCHESS - Identified Patient (IP)
Number analyzed (Participants) | 67 | 66 | 66
percentage of high-risk drinking days
  Baseline | 53.99 (3.03) | 48.14 (3.61) | 41.89 (3.13)
  4 Months | 21.64 (3.43) | 23.98 (4.17) | 22.41 (3.52)
  8 Months | 20.91 (3.54) | 5.49 (4.56) | 4.93 (3.58)
  12 Months | 19.76 (3.62) | 5.92 (4.5) | -7.23 (3.97)

2. Primary Outcome: Psychological Distress
Description: The OQ45 measures the patient's and partner's outcomes during treatment by assessing three sub-domains, Symptom Distress, Interpersonal Relations, and Social Role. Scores from the Outcomes Questionnaire-45 range from 0-180, the higher the score, the higher the symptoms of distress. Cut-off score: 63 or more - indicates symptoms of clinical significance A high score suggests that the client is admitting to a large number of symptoms of distress (mainly anxiety, depression, somatic problems and stress) as well as difficulties in interpersonal relationships, social role (such as work or school), and in their general quality of life. Reliable change: indicated when a client's score changes by 14 points or more.
Time Frame: Baseline, 4, 8, and 12 months
Population: All participants (identified patients and concerned significant others from each arm) were surveyed at baseline, 4, 8, and 12 months.
Measure: Mean (Standard Deviation); unit: score on a scale from 0-180
Arm/Group | Smartphone Control - Identified Patient (IP) | ACHESS - Identified Patient (IP) | PartnerCHESS - Identified Patient (IP) | Smartphone Control - Concerned Significant Other (CSO) | ACHESS - Concerned Significant Other (CSO) | PartnerCHESS - Concerned Significant Other (CSO)
Number analyzed (Participants) | 67 | 66 | 66 | 67 | 66 | 66
score on a scale from 0-180
  Baseline | 69.77 (1.93) | 71.97 (2.28) | 70.35 (1.98) | 51.16 (1.91) | 48.37 (1.87) | 52.85 (1.88)
  4 Months | 69.01 (2.03) | 67.60 (2.41) | 63.89 (2.10) | 51.44 (2.00) | 48.15 (1.94) | 55.01 (1.97)
  8 Months | 63.66 (2.06) | 62.06 (2.50) | 59.17 (2.10) | 51.91 (1.98) | 47.88 (1.94) | 53.85 (2.02)
  12 Months | 63.90 (2.10) | 57.10 (2.51) | 56.64 (2.15) | 53.11 (2.03) | 44.70 (1.91) | 51.86 (1.98)

3. Secondary Outcome: % Days Abstinent
Description: % days abstinent will be measured through the Timeline Followback every 120 days.
Time Frame: Baseline, 4, 8, and 12 months
Population: Identified patients were surveyed at baseline, 4, 8, and 12 months.
Measure: Mean (Standard Deviation); unit: percentage of days abstinent
Arm/Group | Smartphone Control - Identified Patient (IP) | ACHESS - Identified Patient (IP) | PartnerCHESS - Identified Patient (IP)
Number analyzed (Participants) | 67 | 66 | 66
percentage of days abstinent
  Baseline | 26.77 (3.62) | 28.51 (4.33) | 38.61 (3.67)
  4 Months | 55.59 (3.89) | 52.65 (4.84) | 61.20 (4.02)
  8 Months | 59.26 (3.97) | 68.24 (5.11) | 74.65 (3.98)
  12 Months | 65.33 (4.08) | 79.19 (5.14) | 86.59 (4.28)

4. Secondary Outcome: Relationship Satisfaction
Description: Determined by use of the Dyadic Adjustment Scale - 7 (DAS-7) which is a brief version of the 32 question Dyadic Adjustment Scale (DAS) and assesses the quality of marriage and similar dyads. Possible range is 0-36. Higher scores indicate more positive relationship quality. Scores less than 21 are considered to indicate a relationship in distress.
Time Frame: Baseline, 4, 8, and 12 months
Population: Romantic dyads (identified patients and concerned significant others from each arm who stated their partner was a significant other/spouse at baseline) were surveyed at baseline, 4, 8, and 12 months.
Measure: Mean (Standard Deviation); unit: score on a scale from 0-36
Arm/Group | Smartphone Control - Identified Patient (IP) | ACHESS - Identified Patient (IP) | PartnerCHESS - Identified Patient (IP) | Smartphone Control - Concerned Significant Other (CSO) | ACHESS - Concerned Significant Other (CSO) | PartnerCHESS - Concerned Significant Other (CSO)
Number analyzed (Participants) | 44 | 43 | 38 | 45 | 43 | 38
score on a scale from 0-36
  Baseline | 22.87 (.58) | 22.09 (.68) | 22.74 (.63) | 21.66 (.62) | 22.86 (.62) | 23.25 (.69)
  4 Months | 21.66 (.62) | 22.79 (.74) | 21.75 (.67) | 21.48 (.64) | 21.43 (.65) | 21.95 (.72)
  8 Months | 20.89 (.62) | 21.96 (.76) | 20.63 (.66) | 20.36 (.63) | 20.21 (.65) | 22.46 (.73)
  12 Months | 21.98 (.63) | 22.10 (.77) | 20.73 (.68) | 21.90 (.65) | 22.39 (.64) | 22.04 (.72)

ADVERSE EVENTS:
Time Frame: 1 year
Description: Adverse events in Redcap
Arm/Group | Smartphone Control - Identified Patient (IP) | ACHESS - Identified Patient (IP) | PartnerCHESS - Identified Patient (IP) | Smartphone Control - Concerned Significant Other (CSO) | ACHESS - Concerned Significant Other (CSO) | PartnerCHESS - Concerned Significant Other (CSO)
All-Cause Mortality (participants affected / at risk) | 0/67 | 1/66 | 0/66 | 0/67 | 0/66 | 0/66
Serious Adverse Events (participants affected / at risk) | 0/67 | 0/66 | 0/66 | 0/67 | 0/66 | 0/66
Other Adverse Events (participants affected / at risk) | 0/67 | 0/66 | 0/66 | 0/67 | 0/66 | 0/66

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2023-09-07): https://cdn.clinicaltrials.gov/large-docs/28/NCT05419128/Prot_SAP_000.pdf
  • Informed Consent Form: Partner Version (2022-03-30): https://cdn.clinicaltrials.gov/large-docs/28/NCT05419128/ICF_001.pdf
  • Informed Consent Form: Patient Version (2022-03-30): https://cdn.clinicaltrials.gov/large-docs/28/NCT05419128/ICF_002.pdf